CLINICAL TRIAL: NCT04577508
Title: Efficacy of Functional Remediation on Cognitive and Psychosocial Functioning in Patients With Bipolar Disorder: a Randomized Controlled Trial
Brief Title: A Trial of Functional Remediation in Patients With Bipolar Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Antonio Vita, Head Department of Mental Health and Addiction Services, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NP 3976
Record Dates: First submitted 2020-09-30; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Psychosocial Functioning; Functional Remediation; Mood Disorder; Cognitive Enhancement; Cognitive Dysfunctions; Psychosocial interventions; Cognitive Remediation
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders; Cognitive Dysfunction | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Remediation (Experimental): Functional Remediation
  Interventions: Behavioral: Functional Remediation
- Control (Other): Treatment as usual
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Functional Remediation — Functional Remediation is a manualized, group-based psychosocial intervention built on a neurocognitive-behavioural approach, involving modeling techniques, role-playing tasks, self-instruction, positive reinforcement and metacognitive cues (Vieta E et al, Cambridge University Press, 2014). It consists of 21 90-min weekly sessions, in which a trained therapist and co-therapist work with 10-12 patients: the first 3 sessions are dedicated to psychoeducation on neurocognitive deficits; then 13 sessions of neurocognitive training sequentially target attention, memory and executive functions domains, comprising exercises carried out individually, in pairs or in small groups; the last 5 sessions focus on skills training (communication, interpersonal relationships, autonomy, stress management). Content of the sessions involves ecological tasks adapted to real-world situations, and to-be-performed in two contexts (clinical and daily). Homework is assigned, collected and discussed each time.
  Arms: Functional Remediation
Other: Treatment as usual — Standard care for bipolar disorders according to good clinical practice, including drug therapy and individual case management.
  Arms: Control

SUMMARY:
In the last decade several evidences show that cognitive impairment is a major feature of bipolar disorder (BD), that is strongly associated with patients' functional outcome. The most affected cognitive domains in BD are attention, memory and executive functions. BD represents a mental illness of considerable therapeutic complexity and the fight against cognitive and functional deterioration have contributed to increase the interest in the development of specific therapeutic strategies.There is the need of new non-pharmacological interventions in BD in order to improve not only affective symptoms, but also cognitive dysfunctions, with the final goal to achieve full functional recovery. The present study is focused on Functional Remediation (FR), a novel group intervention created by the Bipolar Disorder Unit of the Hospital Clinic of Barcelona and designed specifically for bipolar patients, based on a neuro-cognitive-behavioural approach. It involves neurocognitive and psychoeducation techniques (21 weekly sessions). The present study aims to assess FR efficacy in improving cognitive deficits and psychosocial functioning in a sample of euthymic patients with BD, compared to standard treatment (TAU). This is a randomized and rater-blind trial, involving 54 adult out-patients diagnosed with BD I or II (DSM-5 criteria) and clinically stable for at least two months. Patients will be assessed at baseline, post-treatment and 6-months follow-up, on validated cognitive, clinical and functional rating scales. The main result expected is that patients receiving FR will show better cognitive and psychosocial performance, further confirming the preliminary evidence on the utility of FR as an element of standard care for BD patients.

DETAILED DESCRIPTION:
The main objective of this randomized, rater-blind controlled trial is to evaluate the efficacy of Functional Remediation (FR) in improving functional, clinical and cognitive outcomes in euthymic and clinically stable patients with Bipolar Disorder.

FR is a novel group-based intervention, based on a neurocognitive-behavioural approach, making use of ecological techniques, specifically developed for patients with Bipolar Disorder and aimed at restoring psychosocial functioning in this population.

The study will involve subjects recruited from outpatient clinics (residential or semi-residential care) within the Department of Mental Health and Addiction Services of ASST Spedali Civili, Brescia, Italy.

Study participants will be assigned via central randomization to either FR or treatment as usual, the latter consisting of evidence-based drug treatment and case management.

Pharmacological treatment will be maintained stable during the course of the trial, but no restriction will be applied in terms of access to evidence-based non-pharmacological interventions.

Efficacy of the study intervention (lasting 6 months) will be assessed at post-treatment, and later investigated at 6-months follow-up.

The study will be conducted in accordance with the ethical principles of the Declaration of Helsinki and Good Clinical Practice. It will take place within an experimental project related to the "PhD Course in Biomedical Sciences and Translational Medicine", curriculum "Neuroscience" of the University of Brescia, Italy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of Bipolar Disorder, type I or II, as referred from treating psychiatrist, confirmed at recruitment using the Structured Clinical Interview for Disorder for DSM-5, Clinical Version (SCID-5-CV);
* Clinically stable (in euthymic phase, defined as Y-MRS <= 6 points + HAM-D <= 8 points) for at least 2 months;
* Aged from 18 to 55 years, with no restriction in terms of gender or ethnicity
* With a minimum education level of 8 years;
* Fluent in Italian language;
* Giving written informed consent to study participation.

Exclusion Criteria:

* Intellectual disability (according to DSM-5 criteria);
* Any medical condition that may affect neuropsychological performance (such as neurological diseases);
* Any comorbid psychiatric condition (including current alcohol and/or drug abuse - up to 3 months before screening)
* Pregnancy;
* Inability to provide informed consent/ withdrawal of consent.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Psychosocial functioning | Baseline to post-treatment (6 months)
  Functional outcome will be rated using the Functioning Assessment Short Test (FAST) - Italian Version (Barbato et al., 2013)
Psychosocial functioning | Baseline to follow-up (12 months)
  Functional outcome will be rated using the Functioning Assessment Short Test (FAST) - Italian Version (Barbato et al., 2013)

SECONDARY OUTCOMES:
Neurocognitive performance | Baseline to post-treatment (6 months)
  Neurocognitive performance will be tested using a complete neuropsychological battery specifically developed for patients with bipolar disorder: the Brief Assessment of Cognition in Affective Disorders (BAC-A) (Keefe et al., 2014), Italian normative data (Rossetti et al. 2019)
Neurocognitive performance | Baseline to follow-up (12 months)
  Neurocognitive performance will be tested using a complete neuropsychological battery specifically developed for patients with bipolar disorder: the Brief Assessment of Cognition in Affective Disorders (BAC-A) (Keefe et al., 2014), Italian normative data (Rossetti et al. 2019)
Socio-cognitive performance/Emotional processing | Baseline to post-treatment (6 months)
  Social cognition will be evaluated using the Mayer-Salovey-Caruso Emotional Intelligence Test (MSCEIT), Italian version (Curci et al, 2003)
Socio-cognitive performance/Emotional processing | Baseline to follow-up (12 months)
  Social cognition will be evaluated using the Mayer-Salovey-Caruso Emotional Intelligence Test (MSCEIT), Italian version (Curci et al, 2003)
Subthreshold manic symptoms | Baseline to post-treatment (6 months)
  Manic symptoms will be evaluated using the Young Mania Rating Scale (Y-MRS) (Young et al, 1978). Euthymia will be defined by a score of Y-MRS <= 6 points.
Subthreshold manic symptoms | Baseline to follow-up (12 months)
  Manic symptoms will be evaluated using the Young Mania Rating Scale (Y-MRS) (Young et al, 1978). Euthymia will be defined by a score of Y-MRS <= 6 points.
Subthreshold depressive symptoms | Baseline to post-treatment (6 months)
  Depressive symptoms will be evaluated using the Hamilton Depression Rating Scale (HAM-D) (Hamilton et al, 1960). Euthymia will be defined by a score of HAM-D <= 8 points.
Subthreshold depressive symptoms | Baseline to follow-up (12 months)
  Depressive symptoms will be evaluated using the Hamilton Depression Rating Scale (HAM-D) (Hamilton et al, 1960). Euthymia will be defined by a score of HAM-D <= 8 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Mental Health and Addiction Services, Brescia, BS, Italy

IPD SHARING:
Plan to Share IPD: Undecided